CLINICAL TRIAL: NCT03321630
Title: A Phase II Study of Lenvatinib, a Multi-targeted Tyrosine Kinase Inhibitor, Combined With Pembrolizumab (PD-1 Inhibitor) for the Treatment of Metastatic Gastroesophageal Cancer Patients Who Have Progressed on First or Subsequent Line Therapies
Brief Title: A Phase II a Study of Lenvatinib, a Multi-targeted Tyrosine Kinase Inhibitor, Combined With Pembrolizumab (PD-1 Inhibitor) for the Treatment of Metastatic Gastroesophageal Cancer Patients Who Have Progressed on First or Subsequent Line Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00626; NCT03413397 (obsolete NCT alias)
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: GastroEsophageal Cancer; Gastric Cancer
Keywords: Pebrolizumab; Lenvatinib
MeSH Terms: conditions — Stomach Neoplasms | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenvatinib & Pembrolizumab (Other)
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 20 mg orally each day on days 1-7
Drug: Pembrolizumab — Pembrolizumab 200mg intravenously, to be initiated on day 8, and continued every 3 weeks, in combination with daily lenvatinib 20 mg

SUMMARY:
This is an open label, single arm phase II study, to determine the overall response rate for the combination of lenvatinib and pemrolizumab in patients with metastatic gastroesophageal cancer who have progressed on first or subsequent line therapies. Given the significant cross talk between angiogenesis and the immune response, combined therapy with lenvatinib and pemrolizumab in advanced gastroesophageal cancer patient will provide improved outcomes compared to standard treatment with currently approved agents.

DETAILED DESCRIPTION:
The objective of this study is to determine the progression free survival (PFS), overall survival (OS) and toxicity rates in advanced gastroesophageal patients treated with lenvatinib and pemrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be greater than 18 years of age on day of signing informed consent.
* Have histologically or cytologically confirmed metastatic or recurrent gastric or GEJ adenocarcinoma.
* Have measurable disease based on RECIST 1.1.
* Must have received and have progressed, or are intolerant to at least one systemic regimen (platinum- or fluoropyrimidine-based chemotherapy regimen for metastatic or recurrent disease.)
* If Her2 positive, must have received and have progressed or are intolerant to treatment with trastuzumab for metastatic or recurrent disease.
* Subjects must consent to provide archival tumor tissue (initial and subsequent tumor biopsy samples, if possible) for correlative biomarker studies.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Adequately controlled blood pressure with or without antihypertensive medications defined as BP < 140/90 mmHg at screening and no change in antihypertensive mediation within 1 week prior to the Screening Visit.
* Demonstrate adequate organ function as defined in Table 5, all screening labs should be performed within 10 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential (Section 5.5.2) must be willing to use an adequate method of contraception as outlined in Section 5.5.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.
* Male subjects of childbearing potential (Section 5.5.2) must agree to use an adequate method of contraception as outlined in Section 5.5.2 - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or lenvatinib or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, a minimum of four weeks must have passed and they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Subjects having >1+ proteinuria on urine dipstick testing will undergo 24h urine collection for quantitative assessment of proteinuria. Subjects with urine protein >1g/24h will be ineligible.
* Gastrointestinal malabsorption or any other condition in the opinion of the investigator that might affect the absorption of lenvatinib.
* Prolongation of QTcF interval to >480ms
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug.
* Bleeding disorders or active significant bleeding (i.e. hemoptysis, hematochezia, hematemesis) within 3 weeks.
* Thrombotic disorders or use of anticoagulants, such as warfarin, requiring therapeutic international normalized ratio (INR) monitoring. (treatment with low molecular weight heparin (LMWH) or direct acting oral anti-coagulants is allowed.)
* History of prior gastrointestinal fistula and/or perforation.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Arrhythmias requiring Class Ia and III antiarrhythmics and/or grade >2 bradycardia.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Oberstein, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - The Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenvatinib & Pembrolizumab
Started | 24
Completed | 20
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Investigator Discretion | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenvatinib & Pembrolizumab
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 62 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate as measured by RECIST 1.1; percentage of participants who experience a best overall response of either Complete Response (CR) or Partial Response (PR).
Time Frame: Up to Month 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib & Pembrolizumab
Number analyzed (Participants) | 20
percentage of participants | 25 [8.7 to 49]

2. Primary Outcome: Overall Survival (OS)
Description: Estimated using Kaplan-Meier curve; interval from start of treatment to death due to any cause.
Time Frame: Up to Month 18
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenvatinib & Pembrolizumab
Number analyzed (Participants) | 24
weeks | 21.4 [15.7 to 74.0]

3. Primary Outcome: Progression-Free Survival (PFS)
Description: Estimated using Kaplan-Meier Curves; interval between the date of start of treatment and the earlier date of objective disease progression per RECIST 1.1 criteria or death due to any cause in the absence of progression.
Time Frame: Up to Month 18
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenvatinib & Pembrolizumab
Number analyzed (Participants) | 24
weeks | 12.9 [8.6 to 41.3]

ADVERSE EVENTS:
Time Frame: 18 months
Description: Systematic assessments (regulator investigator assessment at each study visit)
Arm/Group | Lenvatinib & Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 18/24
Serious Adverse Events (participants affected / at risk) | 14/24
Other Adverse Events (participants affected / at risk) | 18/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib & Pembrolizumab (N=24)
Abdominal Pain (Gastrointestinal disorders) | 13
Acute Kidney Injury (Renal and urinary disorders) | 1
Alkaline Phosphatase Increased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Blood Bilirubin Increased (Investigations) | 5
Confusion (Psychiatric disorders) | 2
Death Nos (General disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Gastric Hemorrhage (Gastrointestinal disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Hepatic Failure (Hepatobiliary disorders) | 1
Lung Infection (Infections and infestations) | 1
Renal Colic (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib & Pembrolizumab (N=24)
Abdominal Pain - Right Side (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Agitation (Psychiatric disorders) | 1
Alanine Aminotranferase Increased (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 4
Alk Phosphatase Increased (Investigations) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
ALT increased (Investigations) | 2
Anal Hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthralgia-Knees (Musculoskeletal and connective tissue disorders) | 1
Arthralgias (Musculoskeletal and connective tissue disorders) | 1
Arthralgias B/L Wrists And Knees (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Aspartate Aminotransferase (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 8
Ast Increased (Investigations) | 3
B/L Edema Limbs (General disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Blood Bilirubin Increased (Investigations) | 1
Blurred Vision (Eye disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Bruising-Left Side Of Face (Injury, poisoning and procedural complications) | 1
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1
Chills (General disorders) | 4
Cold Hands (General disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine Increased (Investigations) | 3
Cystitis (Renal and urinary disorders) | 1
Decreased Lymphocyte Counta (Investigations) | 1
Decreased Platelet Count (Investigations) | 1
Decreased White Blood Cells (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 5
Dry Mouth (Gastrointestinal disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Dry Skin - Hands (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Ear Pain (Ear and labyrinth disorders) | 1
Edema Limbs Ankles (General disorders) | 1
Endocrine-Other: Thyroiditis (Endocrine disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Euphoria (Psychiatric disorders) | 1
Fatigue (General disorders) | 13
Fever (General disorders) | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 2
Flank Pain - Left (Musculoskeletal and connective tissue disorders) | 1
Flushing (Vascular disorders) | 1
Gait Disturbance (General disorders) | 1
Gastrointestinal Disorders - Other, Early Satiety (Gastrointestinal disorders) | 1
Gastrointestinal Disorders, Other: Mouth Sores (Gastrointestinal disorders) | 1
Gastrointestinal Disorders- Other: Abdominal Cramping (Gastrointestinal disorders) | 1
General - Others, Blood In Mouth (General disorders) | 1
General - Others, Diaphoresis (General disorders) | 1
General - Others, Hoarse Voice (General disorders) | 1
General - Others, Sweating (General disorders) | 1
General Disorders And Administration Site Conditions - Other, Night Sweats (General disorders) | 1
General Disorders And Administration Site Conditions - Other: Cold Forehead (General disorders) | 1
General Disorders And Administration Site Conditions Other Gum Pain (General disorders) | 1
General Other - Coccyx Pain (General disorders) | 1
General Other - Dark Stool (General disorders) | 1
General Other - Early Satiety (General disorders) | 1
General Other - Gout (General disorders) | 1
General Other - Rhinorrhea (General disorders) | 1
General Other: Chest Redness (General disorders) | 1
Gi Other - Belching (Gastrointestinal disorders) | 1
Gi Other Epigastric Pain (General disorders) | 1
Gi Other: Abdominal Tenderness (Gastrointestinal disorders) | 1
Gum Pain (General disorders) | 1
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 7
Hearing Impaired (Ear and labyrinth disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hyperglycemia Intermittent (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 6
Hypoalbminemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Increased Alkaline Phosphatase (Investigations) | 1
Increased Creatinine (Investigations) | 1
Inr Increased (Investigations) | 2
Insomnia (Psychiatric disorders) | 3
Laryngitis (Infections and infestations) | 1
Left Anterior Thigh Pain (Musculoskeletal and connective tissue disorders) | 1
Left Knee Pain (Musculoskeletal and connective tissue disorders) | 1
Localized Edema (General disorders) | 1
Localized Edema - Legs/Feet (General disorders) | 1
Lower Gum Pain (General disorders) | 1
Lymphocyte Count Decreased (Investigations) | 15
Lymphocyte Count Increased (Investigations) | 2
Mucositis Oral (Gastrointestinal disorders) | 1
Musculoskeletal And Connective Tissue Disorder - Other Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Myalgias (Musculoskeletal and connective tissue disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (General disorders) | 14
Nausea Intermittent (Gastrointestinal disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Nervous System Disorders - Other, Thumb Numbness (Nervous system disorders) | 1
Neutrophil Count Decreased (Investigations) | 3
Oral - Dysesthesia (Nervous system disorders) | 1
Oral Mucositis (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Pain ( Right Neck Pain) (Musculoskeletal and connective tissue disorders) | 1
Pain (Abdominal Pain) (Gastrointestinal disorders) | 1
Pain - Left Hip (Musculoskeletal and connective tissue disorders) | 1
Pain - Left Leg (Musculoskeletal and connective tissue disorders) | 1
Pain - Right Foot (Musculoskeletal and connective tissue disorders) | 1
Pain - Right Leg And Buttock (Musculoskeletal and connective tissue disorders) | 1
Pain In Back Of Head (Nervous system disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Palmar Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodyseshesia Syndrome Intolerable (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2
Palmer Planter Erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1
Palmer-Planter Erythrodysethesia Syndrome (Skin and subcutaneous tissue disorders) | 1
Partial Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Penile Pain (Reproductive system and breast disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Platelet Count Decrease Intermittent (Investigations) | 1
Platelet Count Decreased (Investigations) | 10
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 7
Pruritis (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 3
Rash Maculo Papular (Skin and subcutaneous tissue disorders) | 2
Rash On Face (Skin and subcutaneous tissue disorders) | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Right Knee Pain (Musculoskeletal and connective tissue disorders) | 1
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Skin And Subcutaneous Tissue Disorders - Other, Lesion Under Left Nipple (Skin and subcutaneous tissue disorders) | 1
Skin Hyperpigmentation Black Discoloration Of Feet (Skin and subcutaneous tissue disorders) | 1
Skin Infection (Infections and infestations) | 1
Skin Other Sweating (Skin and subcutaneous tissue disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2
Stomach Pain (Gastrointestinal disorders) | 2
Tachycardia (Cardiac disorders) | 2
Testicular Pain (Reproductive system and breast disorders) | 1
Thromboembolic Event (Vascular disorders) | 2
Tremor In Hands (Nervous system disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Urinary Urgency (Renal and urinary disorders) | 1
Urobilinogenuria (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vaginal Bleeding (Reproductive system and breast disorders) | 1
Vertigo (Nervous system disorders) | 1
Vertigo - Intermittent (Nervous system disorders) | 1
Vomiting Intermittent (Gastrointestinal disorders) | 1
Weight Loss (Investigations) | 5
White Blood Cell Count Decreased (Investigations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT03321630/Prot_SAP_000.pdf